CLINICAL TRIAL: NCT06012305
Title: The Effect of Different KT Applications on Tissue Stiffness, Pain and Function
Brief Title: The Effect of KT on Tissue Parameters
Acronym: KinesioTape
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Nilsah YILMAZ, Lecturer, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GaziosmanpasaU-FTR
Record Dates: First submitted 2023-08-17; First posted 2023-08-25 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Athletic Tape; Trigger Points
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Exercise; Acupressure

STUDY DESIGN:
Intervention Model Description: In the study, there were three groups in which three different treatment programs were applied.
Who Masked: Outcomes Assessor
Masking Description: The person who will make the assessments will not know in which group the individual he/she is assessing is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Only Exercise Group (No Intervention): They will be included in the exercise program that includes postural exercises after ischemic compression and stretching. Stretching exercises will be aimed at stretching the upper trapezius muscle. In the sitting position, the person whose head will be flexed and lateral flexed to the opposite side will stay in this position for 30 seconds and then come back to the same position.
  This will be practiced 15 times a day, 3 days a week. Ischemic compression will then be applied. In ischemic compression, the therapist will apply pressure on the trigger points detected by palpation for 1 minute, and the application will be completed with a total of 5 repetitions at 1-minute intervals. It will continue to be applied 3 sets a day, 3 days a week. Posture exercises were determined as scapular retraction and chin tuck exercises. The exercises will be done in 3 sets of 15 repetitions per day, 3 days a week.
- Taping Group with Muscle Technique (Active Comparator): In addition to the exercise program in the first group, upper trapezius inhibition tape will be applied on the myofascial trigger points in the upper trapezius 3 times a week. The KT (Kinesio Tex Tape, Kinesio Holding Corporation, Albuquerque, USA) used in this study will be waterproof, porous and adhesive. 5 cm wide and 0.5 mm thick kinesio tape will be used. Before the application, the patient will be seated and asked to bring the neck to the opposite side lateral flexion and the head to the same side rotation. In this position, the Kinesiotape inhibition technique will be applied. The tape will be asked to stay on the person for 2 days, then it will be interrupted for 1 day and then the same application will be made. This practice will continue during the 4 weeks of treatment.
  Interventions: Other: Taping
- Taping Group with Epidermis Dermis Fascia Technique (Experimental): In addition to the exercise program in the first group, kinesio taping will be applied with web cut cutting with EDF technique on myofascial trigger points in the upper trapezius. Before the application, the patient will be seated and asked to bring the neck to the opposite side lateral flexion and the head to the same side rotation. Tape will be applied with EDF technique. The band will be asked to stay on the person for 2 days, then a break for 1 day and then the same application will be made again. This practice will continue during the 4 weeks of treatment.
  Interventions: Other: Taping

INTERVENTIONS:
Other: Taping — Taping has the effect of accelerating the flow in the tissue by increasing the epidermal dermal distance. The muscle technique used in the study will be applied to the trapezius muscle and aims to reduce the working level of the muscle. The EDF technique, which will be used in another group, aims to create a stronger base taping effect.
  Other Names: Exercise; ischemic compression
  Arms: Taping Group with Epidermis Dermis Fascia Technique; Taping Group with Muscle Technique

SUMMARY:
Myofascial pain is a concept that refers to pain from trigger points. The region of the upper trapezius muscle is the most common region of myofascial pain syndrome (MAS). It is known that MAS is associated with disruptions in the fascia. It has been observed that kinesio taping supports healing by increasing the epidermal dermal distance. It is thought that the EDF (Epidermis Dermis Fascia) technique provides this effect on the fascia. This idea needs to be put forward with objective data and the study was designed for this purpose. It has been observed that kinesio taping with the inhibition technique for the upper trapezius trigger point has a positive effect on pain and function. Therefore, it will be investigated whether the EDF technique and the inhibition technique have any advantages over each other. An exercise program will be applied to all three groups in the study design, so whether taping provides an additional benefit to fascia smoothness, pain and function will be examined and the 4-week long-term effect of taping, which is mostly short-term effect, will be revealed.

DETAILED DESCRIPTION:
Myofascial pain is a concept that refers to pain from myofascial trigger points. Certain small, hardened, tender areas in the muscle that can be identified by palpation are called trigger points. The upper trapezius is the most common area of myofascial pain syndrome. Working at a desk for a long time and doing intense overhead activities are among the important reasons for this. Individuals who experience myofascial pain with an upper trapezius trigger point are adversely affected in many ways professionally and socially. The pathophysiological process that causes this pain is also related to fascia involvement. It is thought that a taping application that will provide a corrective effect on the fascia will reduce myofascial pain symptoms. The study was designed with the aim of demonstrating that it provides this with objective data.

Kinesio taping increases the epidermal-dermal distance and provides an effect that accelerates the healing after injury. It has been widely preferred in our country and in other countries before, and there is literature support that it can be used safely. It is seen that the inhibition technique is frequently preferred when taping is used in the presence of an upper trapezius trigger point. It is thought that trigger point symptoms will be reduced by inhibiting the upper trapezius muscle to a certain extent with this technique, and some studies in which this effect is achieved are included in the literature. Another taping technique, the Epidermis Dermis Fascia technique (EDF), has been reported to have a healing effect on fascia as clinical opinion, but there is a lack of evidence in the relevant literature.

At the end of the study, the answers to the questions of whether the inhibition technique, which is one of the frequently used techniques, or the epidermis dermis fascia technique, which is at the forefront with its effect on fascia, will be more effective on fascia smoothness, pain and function will be found. With the provision of fascia correction, it is aimed to reduce pain and increase function. It is thought that these gains will reduce the negative effects of myofascial pain.

In addition to taping, two groups will be given an exercise program with proven effect of reducing pain and increasing function in myofascial pain syndrome. The program will include ischemic compression and posture exercises.

The aspects that have not been revealed in previous studies and are considered to be deficiencies are as follows: Which tape technique should be used, which one can be more beneficial? In which of the parameters of pain, function and fascia smoothness will the benefit be valid? What is the long-term effect of kinesio taping, which has a pain-reducing and function-enhancing effect in the short term?

ELIGIBILITY:
Inclusion Criteria:

* Patients with a differential diagnosis of myofascial pain syndrome with unilateral or bilateral active trigger points in the upper trapezius muscle will be included in the study. The criteria for trigger point detection are stated in the literature as follows: 1) The muscle has a challenging palpation area (this area is called the taut band) 2) The trigger point with localized sensitivity in the taut band 3) Typical pain when continuous pressure is applied to the trigger point in the taut band. , numbness, tingling, 4) Local twitching response when the taut band is bent horizontally. Other inclusion criteria are: 18-50 years of age, more than two weeks of symptom duration

Exclusion Criteria:

* Having a diagnosis of fibromyalgia syndrome, diagnosis of psychiatric disorders such as anxiety and depression, radiculopathy symptoms, brachial plexopathy or other nerve entrapments, treatment for myofascial pain syndrome in the last six months, having a malignancy, being pregnant, having an infectious disease, having an inflammatory musculoskeletal system disease have had shoulder or neck surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of fascia stiffness by shear wave elastography | Three measurements at once at the beginning and end of 4 weeks, measurement time 5 minutes per session
  The device provides information on hardness by measuring the velocity of shear waves. The transducer probe of the device will be placed on the tight band in the upper trapezius detected by palpation, and after a comfortable expiration, an image will be taken from the region while the person is sitting. It is planned to take 3 images at 10 second intervals. The acquired image presents both quantitative and qualitative data. Shear modulus values of 10x10 mm square images taken on the trigger point will provide objective data on hardness.

SECONDARY OUTCOMES:
Measurement of pain pressure threshold with an algometer | Three measurements at once at the beginning and end of 4 weeks, measurement time 5 minutes per session
  An analog algometer will be used. The device has a disc-shaped rubber tip with a surface area of exactly 1 cm2. Pressure measurements are expressed in kilograms per square centimeter (kg/cm2). Algometer, metal rod will be perpendicular to the skin surface and the patient will sit; Pressure will be applied to the determined trigger point in 1 kg/second increments. The patient will be instructed to indicate the last point at which pain was perceived. After the dial is set to zero, the process will be repeated 3 times for each patient at 1 minute intervals. The average of three readings will be used for analysis. The dial will show a value between 0 and 22. 0 represents the lowest point of the pain threshold, 22 the highest point.
Pain Assessment with Visual Analog Scale | One measurement at the beginning and end of 4 weeks, 30 seconds measurement time per session
  It will be used in two separate pain evaluations for the upper trapezius region and the pain radiating to the neck and back. 0 will indicate no pain, and ten will show the worst pain the patient has ever experienced. Values will be obtained along a 10 cm Visual Analog Scale line using a ruler marked in centimeters.
Evaluation of upper extremity functions | The questionnaire will be administered at the beginning and end of 4 weeks. The application time of the questionnaire is approximately 5 minutes.
  The short version of the Arm, Shoulder, and Hand Problems Questionnaire(DASH) will be used to make this assessment. DASH is a 30-item questionnaire designed to assess musculoskeletal disorders of the upper extremities. At least 27 questions must be completed for scoring. DASH scores range from 0 to 100, with higher scores indicating a higher level of disability. DASH has been reported to be a valid and reliable tool for evaluating various arm functions. There is information in the literature that Quick DASH, which is its short version, can also provide information about upper extremity function in correlation with DASH. Turkish validity and reliability study was conducted.
Neck Disability Index | The questionnaire will be administered at the beginning and end of 4 weeks. The application time of the questionnaire is approximately 5 minutes.
  Vernon and Mion designed the Neck Disability Index (NDI) to assess how neck pain affects activities of daily living. There is a Turkish validity and reliability study. A score between 0 and 50 points can be obtained from the scale. 0 points means no disability, 50 points means very severe disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Quintner JL, Bove GM, Cohen ML. A critical evaluation of the trigger point phenomenon. Rheumatology (Oxford). 2015 Mar;54(3):392-9. doi: 10.1093/rheumatology/keu471. Epub 2014 Dec 3. PMID 25477053
- [Result] Ertekin E, Kasar ZS, Turkdogan FT. Is early diagnosis of myofascial pain syndrome possible with the detection of latent trigger points by shear wave elastography? Pol J Radiol. 2021 Jul 12;86:e425-e431. doi: 10.5114/pjr.2021.108537. eCollection 2021. PMID 34429789
- [Result] Celiker R, Atalay A, Guven Z. Health-related quality of life in patients with myofascial pain syndrome. Curr Pain Headache Rep. 2010 Oct;14(5):361-6. doi: 10.1007/s11916-010-0141-7. PMID 20690001
- [Result] Kafa N, Citaker S, Omeroglu S, Peker T, Coskun N, Diker S. Effects of kinesiologic taping on epidermal-dermal distance, pain, edema and inflammation after experimentally induced soft tissue trauma. Physiother Theory Pract. 2015;31(8):556-61. doi: 10.3109/09593985.2015.1062943. PMID 26492435
- [Result] Akpinar FM, Sindel D, Ketenci A. Investigation of Effectiveness of Two Different Kinesiotaping Techniques in Myofascial Pain Syndrome: An Open-Label Randomized Clinical Trial. Pain Physician. 2021 Sep;24(6):E721-E731. PMID 34554690
- [Result] Dilek B, Batmaz I, Akif Sariyildiz M, Sahin E, Bulut D, Akalin E, Cevik R, Nas K. Effectiveness of training about kinesiotaping in myofascial pain syndrome: A prospective, single-blind, randomized-controlled study. Turk J Phys Med Rehabil. 2021 Mar 4;67(1):17-24. doi: 10.5606/tftrd.2021.4258. eCollection 2021 Mar. PMID 33948539